CLINICAL TRIAL: NCT02090439
Title: Effectiveness of Silodosin in Medical Expulsive Therapy for Ureteral Pelvic Stone From 4 to 10 mm.
Acronym: SiloMET
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Following difficulties in patient recruitment, we were forced to stop the study prematurely.
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHD 062-13
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2015-11

CONDITIONS: Kidney Stone; Expulsive Medical Therapy
MeSH Terms: conditions — Kidney Calculi | interventions — silodosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard treatment with Silodosin (Experimental): Silodosin
  Interventions: Drug: Silodosin
- standard treatment (No Intervention)

INTERVENTIONS:
Drug: Silodosin
  Arms: standard treatment with Silodosin

SUMMARY:
In the diagnosis of renal colic gallstone , in addition to clinical and biological factors, it is a key : medical imaging. Currently , the French recommendations require at least a couple of Abdomen radiography Without Preparation lying face (ASP ) associated with abdominal ultrasound . "The abdominopelvic CT scan without injection of contrast is the examination of choice.

Current recommendations in the management of gallstone colic simply based on the joint use of analgesics , anti inflammatory drugs and control of water intake .

The mechanism of analgesic action of this treatment is a decrease in the pressure in the cavities by decrease in diuresis and inflammation treatment of ureteral permitting passage of urine . )

The expulsive medical therapy remains under evaluation. The French Association of Urology does not recommend at this time for lack of evidence deemed sufficient.

For foreign companies Urology (EAU , AUA) , the use of calcium channel blockers or alpha blockers in the treatment of symptomatic lower ureteral stones (4 to 10mm ) is recommended (grade 1A) . However, there are less formal studies of their effectiveness .

Investigators wish to demonstrate the effectiveness of alpha in medical expulsive therapy for pelvic stones 4 to 10mm .

ELIGIBILITY:
Inclusion Criteria:

* Men
* Women on oral contraception (for women of childbearing age).
* 18 to 60 years.
* First admission to the episode of renal colic without evidence of complication (afebrile without renal input, negative beta-hCG (women of childbearing age) without severe vomiting without uropathy malformation known underlying balance sheet. ).
* In ability to deliver its consent.
* patient with a single calculation pelvic ureteral 4 to 10 mm cross-sectional diameter, with or without calyx calculations (not obstructive), but other calculation ureter.
* Unique pelvic stone :
* Proven by imaging: helical scan without contrast injection-ASP abdominopelvic.
* Radio-opaque to the ASP.
* More than 3mm and <11mm (4 to 10 mm) of cross-sectional diameter.

Exclusion Criteria:

* Pregnant or lactating women scalable
* No oral contraception
* Contraception by intrauterine device .
* Concurrent infection ( positive urine test strip for Nitrites and / or general signs tanks (T ° C > 38 ° 5 or <36 ° 5 or chills) .
* Renal failure ( Creatinine clearance calculated by Cockcroft and Gault <60 mL / min).
* Single functional kidney .
* Treatment with calcium channel blockers or alpha blockers.
* Recent or upcoming cataract surgery .
* Orthostatic hypotension .
* A history of peptic ulcer disease , liver disease , allergy to paracetamol , the ketoprofen .
* History of stroke , heart disease, diabetes.
* History of allergy to any treatment plans.
* Refusal to enter the protocol.
* Already included in the protocol.
* Medication against -indicated in combination with NSAI (vitamin K ..)
* Hepatic Impairment
* Participation in other biomedical research
* Patients with a history of hypersensitivity such as bronchospasm , asthma, rhinitis , urticaria
* Patients with asthma associated with chronic rhinitis, chronic sinusitis and / or nasal polyposis
* History of gastrointestinal bleeding or perforation during previous treatment with NSAI or history of gastrointestinal diseases such as ulcerative colitis, Crohn's diseases, gastrointestinal bleeding , cerebrovascular bleeding or other bleeding evolving
* Patients receiving treatment associated may increase the risk of ulceration or bleeding (glucocorticoids , selective serotonin reuptake inhibitors and antiplatelet agents such as aspirin )
* Patients with uncontrolled hypertension, congestive heart failure , ischemic heart disease, peripheral arterial disease, and / or a history of stroke (including transient ischemic attack)
* Patients treated with potassium-sparing drugs

Pelvic stone :

* Multiple
* Size < 4 mm or > 10mm
* Radiolucent
* Not formally identified by imaging.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
time to expel kidney stone | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: François LUYCKX, PH, Principal Investigator — CHD Vendée La Roche sur Yon
Locations (2):
- France (2):
  - CH Loire Vendée Océan, Challans
  - Centre hospitalier départemental Vendée, La Roche-sur-Yon